CLINICAL TRIAL: NCT00275340
Title: A Pilot Trial of a Home-Based Peer Support Program After Coronary Artery Bypass Graft Surgery
Brief Title: Cardiac Home Education and Support Trial (CHEST): A Pilot Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Kingston Health Sciences Centre (Other)
Responsible Party: Monica Parry, RN, PhD, CCN(C), University of Toronto
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 15880
Record Dates: First submitted 2006-01-10; First posted 2006-01-11 (Estimated); Results first posted 2009-06-08 (Estimated); Last update posted 2009-06-08 (Estimated); Status verified 2009-04

CONDITIONS: Coronary Artery Disease
Keywords: Pain; Depressive Symptoms; Coronary Artery Bypass; Convalescence; Quality of Life; Human Activities
MeSH Terms: conditions — Coronary Artery Disease; Pain; Depression; Convalescence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Peer Support

SUMMARY:
Coronary artery bypass graft (CABG) surgery is performed more frequently on individuals who are older and sicker than in previous years. Increased patient acuity and reduced hospital length of stays leave individuals ill prepared for their recovery following discharge. Individuals experience pain, functional impairment and depressive symptoms following discharge, which persist for 8 weeks in 50% of individuals. Unrelieved pain, functional decline and depressive symptoms predispose individuals to adverse events, impaired health-related quality of life (HRQOL), and increased morbidity and mortality.

Existing supports; including printed education materials, community care resources, cardiac rehabilitation programs and nurse-initiated telephone follow-up, fail to address concerns of individuals in this early period following hospital discharge.

Despite the positive health outcomes in other patient populations, valid studies examining the impact of telephone-based peer support to men and women after hospital discharge from CABG surgery were not found. It is anticipated that a home-based peer support program, delivered by telephone, will improve recovery and enhance HRQOL for individuals in the early weeks post hospital discharge from CABG surgery.

DETAILED DESCRIPTION:
Coronary artery bypass graft (CABG) surgery is performed more frequently on individuals who are older and sicker than in previous years. This, combined with reduced hospital length of stays, leaves individuals ill prepared for their recovery after discharge. Individuals experience pain, functional impairment and depressive symptoms; which predispose them to adverse events and impaired health-related quality of life (HRQOL). A home-based peer support program may improve recovery outcomes for individuals following CABG surgery.

The objectives of this pilot trial were to test the feasibility of all procedures, specifically to determine: 1) an estimate of patient and peer recruitment rates, 2) peer compliance and dose of the intervention, 3) peer satisfaction with orientation, 4) peer support activities offered to patients, and 5) patients' satisfaction with peer support. Additionally, exploratory research questions were used to determine indicators of the effects of peer support on HRQOL, pain, pain-related interference with activities, function, depressive symptoms, and enrolment in cardiac rehabilitation. An 8-week pre-post test RCT design enrolled men and women undergoing CABG surgery at a single site in Southeastern Ontario. Patients were randomized to either a usual care or an intervention group. Patients allocated to usual care received preoperative/postoperative education sessions, a preoperative video/information booklet, and preoperative/postoperative visits from in-hospital peer volunteers. In addition to usual care, patients in the intervention group received individualized education and support via telephone for 8 weeks following hospital discharge from trained peer volunteers.

Peer volunteers participated in a 4-hour orientation session. Ninety-three percent of the peers felt adequately prepared for their peer volunteer role and 98% of them initiated calls within 72 hours of the patient's discharge. Peers made an average of 12 calls, less than 30 minutes in duration, to each patient over the 8-week period. Most common support activities provided by the peers included listening to patient concerns, promoting activities, reinforcing rest periods and encouraging achievements. Patients were satisfied with their peer support experience. The intervention group reported improved physical function, role function, less pain and improved cardiac rehabilitation enrolment.

The evidence obtained from this pilot trial suggests that a home-based peer support intervention is feasible following CABG surgery. The information will be used to plan a larger multi-centre trial.

ELIGIBILITY:
Inclusion Criteria (patients): Men and women who

* are having first-time non-emergency CABG surgery
* are judged ready for discharge
* are being discharged to home [either their own or to family/friends]
* have access to and are able to communicate over a telephone
* are able to read, write and understand English

Inclusion Criteria (peers): Men and women who

* have undergone CABG surgery within the last 5 years
* have access to and are able to communicate clearly over a telephone
* are able to read, write and understand English
* have attended a formal cardiac rehabilitation program
* are not associated with the current in-hospital peer volunteer program

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2006-02; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Monica J. Parry, PhD, Principal Investigator — Faculty of Nursing, University of Toronto
Locations (1):
- University of Toronto, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Parry M, Arthur H, Brooks D, Groll D, Pavlov A. Measuring function in older adults with co-morbid illnesses who are undergoing coronary artery bypass graft (CABG) surgery. Arch Gerontol Geriatr. 2012 May-Jun;54(3):477-83. doi: 10.1016/j.archger.2011.04.013. Epub 2011 Jun 29. PMID 21719124
- [Derived] Parry MJ, Watt-Watson J, Hodnett E, Tranmer J, Dennis CL, Brooks D. Cardiac Home Education and Support Trial (CHEST): a pilot study. Can J Cardiol. 2009 Dec;25(12):e393-8. doi: 10.1016/s0828-282x(09)70531-8. PMID 19960132

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients (n=106) were recruited between April-February 2007. Patients having elective coronary artery bypass graft surgery were recruited at the outpatient preadmission class; those having urgent/semi-urgent surgery were recruited in hospital. Peers (n=20) were recruited from the region of Southeastern Ontario during February-March 2006.
Pre-assignment Details: One hundred and one patients were randomized at hospital discharge to either usual care or peer support. Five patients who were recruited preoperatively did not meet the eligibility criteria postoperatively for randomization. Of the 20 peers recruited, 6 were unable to participate in one of the training sessions offered in April 2006.
Groups:
- Usual Care: Patients allocated to usual care received the standard education/support offered to patients post coronary artery bypass graft surgery: preoperative/postoperative group education, preoperative video, general information booklet and preoperative/postoperative visits from in-hospital peer volunteers.
- Peer Support: In addition to usual care, patients randomly assigned to peer support received individualized pain management and exercise education via home-based peer support delivered by telephone.
Period: Overall Study
Arm/Group | Usual Care | Peer Support
Started | 52 | 49
Completed | 50 | 45
Not Completed | 2 | 4
Not completed — Lost to Follow-up | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Peer Support | Total
Number analyzed (Participants) | 52 | 49 | 101
Age Continuous [Mean (Standard Deviation); unit: years] | 64 (10) | 62 (11) | 64 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 43 | 41 | 84
Left Ventricular Function [Number; unit: Participants]
  Grade 1 (normal) | 32 | 20 | 52
  Grade 2 | 15 | 24 | 39
  Grade 3 | 4 | 5 | 9
  Grade 4 (worst) | 0 | 0 | 0
  No Response | 1 | 0 | 1
Marital Status [Number; unit: participants]
  Married | 38 | 42 | 80
  Divorced/Widow/Single | 13 | 7 | 20
  No Response | 1 | 0 | 1
Health-Related Quality of Life (SF-36v2-Acute Form) [Mean (Standard Deviation); unit: units on a scale] — The SF-36v2 yields a score for each domain of health. All domains are scored on a scale from 0 (negative health) to 100 (positive health), with 100 representing the best possible health state.
  units on a scale
    Physical Function | 57.0 (27.7) | 54.4 (31.7) | 54.7 (29.8)
    Role-Physical | 44.3 (32.4) | 37.6 (30.8) | 40.3 (31.6)
    Bodily Pain | 64.4 (29.0) | 70.4 (25.9) | 67.1 (27.7)
    General Health | 65.3 (18.8) | 64.1 (21.5) | 64.6 (19.8)
    Physical Component Score | 41.2 (11.0) | 40.5 (11.3) | 40.6 (11.1)

OUTCOME MEASURES:

1. Primary Outcome: Health-related Quality of Life (SF-36v2-acute Form)
Description: The SF-36v2 yields a score for each domain of health. All domains are scored on a scale from 0 (negative health) to 100 (positive health), with 100 representing the best possible health state.
Time Frame: 9 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Peer Support
Number analyzed (Participants) | 50 | 45
units on a scale
  Physical Functioning | 72.6 (22) | 77.0 (19.0)
  Role-Physical | 60.4 (29.2) | 65.5 (27.6)
  Bodily Pain | 72.2 (25.7) | 78.8 (21.5)
  General Health | 68.5 (19.5) | 72.2 (17.3)
  Physical Component Summary Scale | 44.6 (9.2) | 47.5 (8.2)
Statistical Analysis 1: Comparison: Usual Care vs Peer Support; Mean change scores were computed on domain and summary scores. Mean differences in change scores between groups were computed and t-tests used to detect significant differences; Test type: Non-Inferiority or Equivalence — Study was not powered to determine significant group differences; thus trends are reported for p<0.20; p < 0.20, t-test, 2 sided

2. Secondary Outcome: Pain (McGill Pain Questionnaire-Short Form)
Time Frame: 9 weeks
Reporting Status: Not Posted, anticipated posting 2009-09
Measure: Number; unit: Participants

3. Secondary Outcome: Interference With Activities (Brief Pain Inventory-Interference Subscale)
Time Frame: 9 weeks
Reporting Status: Not Posted, anticipated posting 2009-09
Measure: Number; unit: participants

4. Secondary Outcome: Function (Human Activity Profile)
Time Frame: 9 weeks
Reporting Status: Not Posted, anticipated posting 2009-09
Measure: Mean (Standard Deviation); unit: participants

5. Secondary Outcome: Depressive Symptoms (Center for Epidemiologic Studies Depression Scale)
Time Frame: 9 weeks
Reporting Status: Not Posted, anticipated posting 2009-09
Measure: Number; unit: participants

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No